CLINICAL TRIAL: NCT02309047
Title: The Cycle Disturbances, OLigomenorrhea and Amenorrhea (COLA) Study & Biobank
Acronym: COLA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Bart CJM Fauser, professor BCJM Fauser, UMC Utrecht
Other Study IDs: 12-645
Record Dates: First submitted 2014-11-12; First posted 2014-12-05 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Anovulation
MeSH Terms: conditions — Anovulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 6 x 500 μL serum, 2 x 500 μL EDTAplasma en 3 x 900 μL celpellet
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- WHO anovulation: WHO I, II. III anovulation. See inclusion criteria

SUMMARY:
Through the COLA Study and Biobank the investigators hope to enable further identification of phenotype, endocrine, ethnic, and metabolic characteristics associated with menstrual cycle disturbances; and: the identification of genetic or other etiologic factors associated with cycle disturbances.

DETAILED DESCRIPTION:
Population Women with cycle disturbances are referred to the outpatient clinic specialized in cycle disturbances by 1st or 2nd line care providers for further diagnostic procedures.

Inclusion criteria WHO I Hypogonadotropic hypoestrogenic status (previously: "hypothalamic amenorrhea")

1. Low to normal serum follicle-stimulating hormone (FSH) concentrations
2. Low serum estradiol concentrations

WHO II

1. Amenorrhea or oligomenorrhea (mean cycle >35 days during the last 6 months)
2. Normal serum FSH concentrations (<12 IU/L)
3. Absence of other causes for the cycle disturbance, including: normal prolactin concentrations (<1.0 IU/L), normal thyroid stimulating hormone (TSH) concentrations (0.2 - 4.2 milli-International unit /L), abnormalities on ultrasonography.

Within women with WHO II status, polycystic ovary syndrome (PCOS) is diagnosed when at least 2 of the following criteria are met:

1. Oligo-/anovulation
2. Clinical and/ or biochemical hyperandrogenism
3. Polycystic ovaries on ultrasonography

WHO III

1. primary ovarian insufficiency (POI): defined as secondary amenorrhea before the age of 40 years and basal FSH > 40 IU/L.
2. incipient ovarian failure (IOF): defined as normal-ovulatory cycles with raised basal FSH > 12 IU/L before the age of 40 years.
3. transient ovarian failure (TOF): defined as irregular cycles with raised basal FSH > 12 IU/L before the age of 40 years.
4. Poor ovarian response: defined as less than 4 oocytes retrieved or cancellation in case of absent follicle growth after ovarian hyperstimulation with 300 IU gonadotropins.
5. Early menopause: menopause occurring between age 40 and 45 years.
6. Hypergonadotropic primary amenorrhea: primary amenorrhea with raised basal FSH > 12 IU/L. Controls For analyses in which comparison with female controls are needed, data will be collected from existing population based cohorts, such as the EPIC cohort (Julius Center), or selected women included in the preconceptional cohort (PC, derived from the Department of Reproductive Medicine and Gynaecology in the University Medical Center Utrecht (UMCU), separate protocol in preparation).

Exclusion criteria

* Age: younger than 18 yrs.
* Regularly cycling women, with the exception of women with elevated basal FSH concentrations (IOF cases).

Study parameters In order to determine the phenotype characteristics of women with cycle disturbances, and to allow for the identification of genetic factors associated with cycle disturbances, the following parameters will be obtained.

* Age
* Ethnicity
* Social economic status and education
* Intoxications: smoking habits (previous and current), use of alcohol or drugs
* Medication and medication history
* Mental health (depression, stress and anxiety)
* Cycle regularity: age at menarche, use of (oral/intrauterine) contraceptives, mean duration of cycle, variation in cycle duration.
* Reproductive & obstetric history: parity, time to pregnancy and pregnancy outcome, subfertility (including treatments)
* Medical history (including previous gonadotoxic treatment)
* Family history of diabetes mellitus, early menopause, cycle irregularities, subfertility, cardiovascular disease, endocrinological disease, congenital disorders
* Basic physical examination: systolic and diastolic blood pressure, height, weight (BMI), waist circumference, hip circumference
* Assessment of hirsutism, acne, Tanner sexual development stages.
* Ovarian reserve parameters: antral follicle count, ovarian volume, anti-müllerian hormone (AMH)
* luteinizing hormone (LH), FSH, prolactin, TSH, estradiol concentrations
* Androgen levels
* Lipid spectrum, glucose, insulin, High sensitivity C-reactive protein
* In POI specifically: bone density as assessed by dual-energy X-ray absorptiometry (DEXA), karyotype, fragile X premutation screening, presence of autoantibodies (against thyroid, ovaries, parietal cells and adrenal gland).

Participation in the COLA Biobank will consist of the additional withdrawal of two blood vials (one for DNA and one for serum sampling) obtained during the routine diagnostic procedure.

Relatives of the index patient:

When a familial tendency of the WHO status is suspected on the basis of family history of 1st and 2nd degree relatives, these relatives will be invited for participation of the study.

ELIGIBILITY:
Inclusion Criteria:

WHO I Hypogonadotropic hypoestrogenic status (previously: "hypothalamic amenorrhea")

1. Low to normal serum FSH concentrations
2. Low serum estradiol concentrations

WHO II

1. Amenorrhea or oligomenorrhea (mean cycle >35 days during the last 6 months)
2. Normal serum FSH concentrations (<12 IU/L)
3. Absence of other causes for the cycle disturbance, including: normal prolactin concentrations (<1.0 IU/L), normal TSH concentrations (0.2 - 4.2 milliunits/L), abnormalities on ultrasonography.

Within women with WHO II status, PCOS is diagnosed when at least 2 of the following criteria are met:

1. Oligo-/anovulation
2. Clinical and/ or biochemical hyperandrogenism
3. Polycystic ovaries on ultrasonography

WHO III

1. POI: defined as secondary amenorrhea before the age of 40 years and basal FSH > 40 IU/L.
2. IOF: defined as normal ovulatory cycles with raised basal FSH > 12 IU/L before the age of 40 years.
3. TOF: defined as irregular cycles with raised basal FSH > 12 IU/L before the age of 40 years.
4. Poor ovarian response: defined as less than 4 oocytes retrieved or cancellation in case of absent follicle growth after ovarian hyperstimulation with 300 IU gonadotropins.
5. Early menopause: menopause occurring between age 40 and 45 years.
6. Hypergonadotropic primary amenorrhea: primary amenorrhea with raised basal FSH > 12 IU/L.

Exclusion criteria: Exclusion criteria

* Age: younger than 18 yrs.
* Regularly cycling women, with the exception of women with elevated basal FSH concentrations (IOF cases).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with cycle disturbances are referred to the outpatient clinic specialized in cycle disturbances by 1st or 2nd line care providers for further diagnostic procedures.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2004-10 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
hormonal classification | within 6 weeks
  FSH, LH, Estradiol, Progesterone,Testosterone, Androstenedione, Sex hormone binding globulin (SHBG), Cortisol, TSH
metabolic profile | within 6 weeks
  total cholesterol, triglycerides, LDL cholesterol, HDL cholesterol, insulin, glucose
ovarian reserve | within 6 weeks
  anti mullerian hormone, FSH and antral follicle count.

SECONDARY OUTCOMES:
autoimmunity in WHO 3- POI patients | within 3 months
  antithyroid peroxidase, antiadrenal, antiparietal and antiovarian antibodies
bone density in WHO 3- POI patients | within 3 months
  a dual-energy x-ray absorptiometry (DEXA) scan
genotype in WHO 3 POI patients | within 3 months
  karotype, fragile X mental retardation 1 gene premutation carriership

CONTACTS AND LOCATIONS:
Overall Officials: Bart CJ Fauser, professor, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Christ JP, Gunning MN, Meun C, Eijkemans MJC, van Rijn BB, Bonsel GJ, Laven JSE, Fauser BCJM. Pre-Conception Characteristics Predict Obstetrical and Neonatal Outcomes in Women With Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2019 Mar 1;104(3):809-818. doi: 10.1210/jc.2018-01787. PMID 30590587
- [Derived] Christ JP, Gunning MN, Palla G, Eijkemans MJC, Lambalk CB, Laven JSE, Fauser BCJM. Estrogen deprivation and cardiovascular disease risk in primary ovarian insufficiency. Fertil Steril. 2018 Apr;109(4):594-600.e1. doi: 10.1016/j.fertnstert.2017.11.035. Epub 2018 Mar 28. PMID 29605405
- See also: study information — https://www.umcutrecht.nl/nl/ziekenhuis/onderzoek/cola-screening